CLINICAL TRIAL: NCT05005117
Title: Laparoscopic Approach for Emergency Colon Resection: a Randomized Controlled Trial
Brief Title: Laparoscopic Approach for Emergency Colon Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Kanta-Häme Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q048
Record Dates: First submitted 2021-07-30; First posted 2021-08-13 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopic Surgery; Colorectal Cancer; Colorectal Disorders; Emergencies; Complication of Surgical Procedure; Long-term Effects of Cancer Treatment
Keywords: Laparoscopic surgery; Emergency surgery; Colorectal
MeSH Terms: conditions — Colorectal Neoplasms; Emergencies | interventions — Heller Myotomy

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled multicenter trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic operation (Experimental): Laparoscopic emergency colon resection
  Interventions: Procedure: Laparoscopic operation
- Open operation (Active Comparator): Open emergency colon resection
  Interventions: Procedure: Open operation

INTERVENTIONS:
Procedure: Laparoscopic operation — Operation
  Arms: Laparoscopic operation
Procedure: Open operation — Operation
  Arms: Open operation

SUMMARY:
This is a randomized, controlled, parallel, multicenter trial to compare post-operative complications and long-term results between open and laparoscopic technique in emergency colorectal surgery.

DETAILED DESCRIPTION:
Laparoscopic technique in elective colorectal surgery has been shown to be advantageous for patients compared to open technique. However, the feasibility and potential benefits of laparoscopic colorectal surgery in emergency setting has not been evaluated sufficiently.

The aim of this study is to compare laparoscopic and open technique in emergency colon resections. Primary outcome is the immediate recovery after operation and secondary outcome is long-term overall and cancer-specific survival.

ELIGIBILITY:
Inclusion Criteria:

* all patients in need of emergency colon resection

Exclusion Criteria:

* age < 18 year
* trauma patients
* reoperations
* acute pancreatitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2031-07-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
postoperative morbidity | 30 days
  Postoperative morbidity evaluated by Clavien-Dindo classification

SECONDARY OUTCOMES:
Surgical site infections | 30 days
  Surgical site infections, superficial and deep
Long-term Survival | 5 years
  Long-term overall and cancer-specific survival

CONTACTS AND LOCATIONS:
Overall Officials: Marie T Grönroos-Korhonen, MD, Principal Investigator — Päijät Häme Central Hospital
Locations (1):
- Marie Grönroos-Korhonen, Lahti, Finland

REFERENCES:
- [Derived] Gronroos-Korhonen MT, Kossi JAO. LapEmerge trial: study protocol for a laparoscopic approach for emergency colon resection-a multicenter, open label, randomized controlled trial. Trials. 2024 Apr 17;25(1):268. doi: 10.1186/s13063-024-08058-0. PMID 38632602